CLINICAL TRIAL: NCT03805880
Title: Cerebral Desaturation During One Lung-ventilation and Postoperative Dysfunction Afterthoracic Surgery: a Prospective Observational Study
Brief Title: Cerebral Desaturation and Postoperative Dysfunction After Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Silvia Fiorelli, principal investigator, University of Roma La Sapienza
Other Study IDs: SATURIMETRIA
Record Dates: First submitted 2019-01-10; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Thoracic Surgery; Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: cerebral desaturation monitoring and cognitive examination — Before general anesthesia, continuous monitoring of cerebral oxygenation(rSO2) was started using an INVOS 5100 (Somaneic, Tro, MI) .Patient cognitive function was assessed using Mini-Mental State Examination (MMSE) on the day before surgery (baseline) and then after 1 day after surgery.

SUMMARY:
The purpose of this study prospective observational study is to determine cognitive dysfunction incidence after thoracic surgery. We also evaluate evaluate the role of cerebral oxygen desaturations and hypertension as risk factors for post-operative cognitive dysfunction (POCD) in patients undergoing lung resection.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective lobectomy or wedge resection via thoracotomy
* one lung ventilation (OLV duration) ≥ 45 min

Exclusion Criteria:

* previous cerebral disease,
* dementia,
* severe cognitive dysfunction
* emergency surgery
* pregnancy
* patient refusal to give consent
* inability to give consent
* age ≤18 years
* ASA ≥ IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for elective lobectomy or wedge resection via thoracotomy requiring an OLV duration ≥ 45 min
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
incidence of cognitive dysfunction after thoracic surgery | change of MMSE score from the day before surgery (baseline) at 1 day after surgery
  A decrease in Mini-Mental State Examination (MMSE) score > 2 points from baseline was defined as Postoperative cognitive dysfunction (POCD)

SECONDARY OUTCOMES:
role of cerebral oxygen desaturations as risk factors for POCD in patients undergoing lung resection. | change of cerebral saturation from baseline(before surgery) at intraoperative measure
  monitoring values of cerebral saturation during intraoperative period:Cerebral desaturation was defined as a reduction of rSO2 during OLV of more than 20% from the baseline value
role of hypertension as risk factors for POCD in patients undergoing lung resection. | change of blood pressure from baseline(before surgery) at intraoperative measure
  monitoring values of blood pressure during intraoperative period

CONTACTS AND LOCATIONS:
Locations (1):
- azienda ospedaliero universitaria Sant'Andrea, Roma, Italy

IPD SHARING:
Plan to Share IPD: No